CLINICAL TRIAL: NCT01628432
Title: Effect of Total Salpingectomy During Conservative Hysterectomy for Benign Disease on Ovarian Function: Non Inferiority Randomized Controlled Trial
Brief Title: Effect of Salpingectomy During Conservative Hysterectomy
Acronym: SALPINGOVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRN11/LO/SALPINGOVA
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Genital Diseases, Female; Hysterotomy; Affecting Fetus; Leiomyomata Uteri; Adenomyosis, Endometriosis; Dysfunctional Uterine Bleeding; Cervical Dysplasia; Uterine Prolapse
MeSH Terms: conditions — Genital Diseases, Female; Adenomyosis; Endometriosis; Metrorrhagia; Uterine Cervical Dysplasia; Uterine Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- conservative hysterectomy I (Experimental): bilateral salpingectomy during hysterectomy with conservation of the ovaries
  Interventions: Procedure: conservative hysterectomy I
- conservative hysterectomy II (Active Comparator): standard conservative hysterectomy with conservation of both ovaries and tubes
  Interventions: Procedure: Conservative hysterectomy II

INTERVENTIONS:
Procedure: conservative hysterectomy I — conservative hysterectomy for benign disease
  Arms: conservative hysterectomy I
Procedure: Conservative hysterectomy II — bilateral salpingectomy during hysterectomy without conservation of the ovaries
  Arms: conservative hysterectomy II

SUMMARY:
The study compares the effect of bilateral salpingectomy associated with conservative hysterectomy on ovarian function to the standard hysterectomy with conservation of both ovaries and tubes in terms of hormone assays, ovarian ultrasound evaluation, complications, quality of life.

DETAILED DESCRIPTION:
Hysterectomy is one of the most common gynecologic procedures performed in clinical practice. In this study we focused on non menopausal patients under 52 years having hysterectomies for benign disease : uterine leiomyomas, adenomyosis, endometriosis, dysfunctional uterine bleeding, genital prolapse, cervical dysplasia... with failure of conservative treatment.

the standard procedure during hysterectomy with conservation of the ovaries has been the preservation of fallopian tubes with the clamps placed as close to the uterine corpus as possible. this is suggested to decrease interference with the vascular structures in the mesosalpinx and mesovarium. however it is unclear whether tubal conservation at the time of hysterectomy has any influence on ovarian blood flow or ovarian reserve. another point to be considered is the occurrence of post-hysterectomy carcinoma in the preserved fallopian tube, theoretically, these cases could be prevented if tubal excision is performed during hysterectomy The study compares the effect of bilateral salpingectomy associated with conservative hysterectomy on ovarian function to the standard hysterectomy with conservation of both ovaries and tubes in terms of hormone assays, ovarian ultrasound evaluation, complications, quality of life.

impact of treatments on ovarian reserve are tested by measuring AMH at baseline and 3 days, 6 weeks and 6, 12 months after surgeries.

quality of life is also assessed at these time points, with a questionnaire (Women Health Questionnaire WHQ).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years and less than 52 years
* indication of a conservative hysterectomy for benign disease
* signed informed consent
* non menopausal women (AMH >0,21 ng/ml)

Exclusion Criteria:

* pregnancy
* desire of future pregnancy
* menopausal status
* patient unable to give informed consent
* any physical or psychiatric condition that could impair with patient's ability to cooperate with post operative data collection
* previous salpingo and /or oophorectomy (unilateral or bilateral)
* genital cancer disease or atypical endometrial hyperplasia
* hyperandrogenia
* any ovarian mass that needs surgical exploration
* any immunotherapy that could interfere with immunological tests

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2012-07; Primary Completion 2017-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
percentage of patients with more than 20% diminution of AMH logarithm at one year (12 months) | one year

SECONDARY OUTCOMES:
AMH measurement at 3 days, 6 weeks, and 6, 12 months after hysterectomy endovaginal ultrasound evaluation of the ovarian volume and vascularisation quality of life (WHQ questionnaire) reintervention procedures complications | day3, week 6, month 6 and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Lobna OULDAMER, MD, Principal Investigator — CHRU de TOURS
Locations (7):
- France (7):
  - CHU, Angers
  - CHU, Le Kremlin-Bicêtre
  - CHU, Lille
  - Hôpital Sud, Lyon
  - CHU, Poitiers
  - CHU, Rennes
  - CHU, Tours